CLINICAL TRIAL: NCT06344026
Title: Phase 1/2a Dose Escalation Study of ANPD001 in Sporadic Parkinson Disease
Brief Title: Phase 1/2a Study of ANPD001 in Parkinson Disease
Acronym: ASPIRO
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Aspen Neuroscience (Industry)
Collaborators: California Institute for Regenerative Medicine (CIRM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANPD001-02
Record Dates: First submitted 2024-03-18; First posted 2024-04-03 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Autologous; Induced Pluripotent Stem Cells; Cell Therapy; Dopamine; Regenerative Medicine
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Open label, dose escalation of bilateral injection of ANPD001 dopaminergic precursor cells to the putamen
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (1):
- ANPD001 (Experimental)
  Interventions: Biological: ANPD001; Device: Custom Device

INTERVENTIONS:
Biological: ANPD001 — Biologic: ANPD001 is an experimental product derived from the patient's own skin cells converted to induced pluripotent stem cells. The stem cells were differentiated into precursors for brain cells that produce dopamine.
Device: Custom Device — A custom device to facilitate slow injection of small volumes of investigational drugs (including cell therapies), under MRI guidance

SUMMARY:
This clinical trial is designed to test the safety and tolerability of injecting ANPD001 cells that will mature into dopamine-producing cells into the brain of participants with Parkinson Disease. All participants will have ANPD001 cells manufactured from their own previously collected cells.

DETAILED DESCRIPTION:
Participants will undergo a surgical implantation of cells that will mature into dopamine-producing neurons under general anesthesia into a part of the brain where dopamine production is decreased in patients with Parkinson Disease. The effect on Parkinson Disease symptoms, safety and tolerability, and cell survival are assessed for 5 years post-transplant (with MRI and PET imaging scans of the brain). Safety and tolerability are assessed annually for an additional 10 years via telephone call (total follow-up of 15 years)

ELIGIBILITY:
Inclusion Criteria:

* Age 50-70 years of age at time of consent in the trial-ready cohort study ANPD001-01
* Met all eligibility requirements for inclusion in the trial-ready cohort in clinical study ANPD001-01
* Diagnosed with Parkinson Disease at least 4 years ago
* Unequivocal motor response to Levodopa

Exclusion Criteria:

* Prior brain surgery that, in the opinion of the neurologist or neurosurgeon, contraindicates administration of ANPD001
* History of intracranial therapy for PD, including deep brain stimulation (DBS), focused ultrasound (FUS), gene therapy or other biological therapy
* History of cognitive impairment or dementia
* History of clinically significant Dopa Dysregulation syndrome
* History of epilepsy, stroke, multiple sclerosis, poorly controlled or progressive neurological disease (other than PD), or poorly controlled cardiovascular disease
* Inability to temporarily stop anticoagulation or antiplatelet therapy for at least 2 weeks
* History of malignancy (cerebral or systemic) within the prior 5 years, except treated cutaneous squamous or basal cell carcinomas
* Contraindication to MRI and/or use of gadolinium
* Weight > 300 lbs or Body Mass Index (BMI) > 35
* Uncontrolled diabetes (HbA1c > 7.0%) or any other acute or chronic medical condition that would significantly increase the risks of a neurosurgical procedure
* Pregnancy or lactation
* Significant drug-induced dyskinesia (>2 for any body part on the Abnormal Involuntary Movement Scale [AIMS])
* Male or female with reproductive capacity who is unwilling to use barrier contraception for 3 months post-administration of the investigational product
* Unable to comply with the protocol procedures, including frequent and prolonged follow-up assessments
* Any significant issue raised by the neurologist or neurosurgeon

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2024-01-23 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2030-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment emergent adverse events (Safety and Tolerability) | 1 year (primary follow up)
  incidence and severity of treatment emergent adverse events (TEAE) and serious adverse events (SAE)

SECONDARY OUTCOMES:
"ON" time without troublesome dyskinesia | 1 year (primary follow up) and 5 years (long term follow up)
Post-injection change in Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II (Activities of Daily Living - ADL) and Part III (motor score) in the ON state (total score and scores for Parts I-IV) | 1 year (primary follow up) and 5 years (long term follow up)
  Part II score range is 0 to 52 with 0 being normal and 30 and above being severe
Post-injection change in the Movement Disorder Society - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III score in the practically defined OFF state | 1 year (primary follow up) and 5 years (long term follow up)
  Part III score range is 0 to 132 with 0 being normal and 59 and above being severe
Post-injection change in the 18F-DOPA uptake in the putamen | 1 year (primary follow up) and 5 years (long term follow up)
  Post-injection change in the 18-fluorodopa uptake in the putamen from baseline via positron emission tomography (PET)
Incidence and severity of treatment emergent adverse events during long term follow-up (Continued Safety and Tolerability) | 14 years of long term follow up (4 years in-person visits and 10 additional years follow up via telephone call)

CONTACTS AND LOCATIONS:
Overall Officials: Edward D Wirth III, MD, PhD, Study Chair — Aspen Neuroscience
Locations (9):
- United States (9):
  - University of Arizona - Banner Health, Tucson, Arizona
  - Scripps Health, La Jolla, California
  - University of California, Los Angeles, Los Angeles, California
  - University of California, Irvine, Orange, California
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - University of Colorado, Aurora, Colorado
  - Emory University, Atlanta, Georgia
  - Feinstein Institutes, Manhasset, New York

IPD SHARING:
Plan to Share IPD: No